CLINICAL TRIAL: NCT06375941
Title: Prospective Observational Study of Localized Angiosarcoma of Any Site: ProStars
Acronym: ProStars
Status: Recruiting | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Other Study IDs: ProStars
Record Dates: First submitted 2024-04-05; First posted 2024-04-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pathological diagnosis of AS, any site of origin, any age, primary, localized, resectable disease.: * pathological diagnosis of AS;
  * any site of origin;
  * any age;
  * primary, localized, resectable disease.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
This study will be a multi-institutional, prospective, observational study of patients with localized primary AS of any site within ISG and RTR centers. Patients will be treated according to clinical practice of the center and according to ISG clinical recommendations on localized AS.

DETAILED DESCRIPTION:
The management of localized AS remains a clinical challenge and needs to be better defined and standardized, especially with regards to the role of radiation-therapy and systemic treatment. Several questions about the best treatment approach to some clinical presentations remain open and would need to be answered by clinical studies. Unfortunately, the rarity of this histology among sarcomas makes it challenging to carry out clinical studies in all such presentations. Moreover, prognostic factors are lacking and differences in epidemiological, pathological and clinical aspects between primary AS and secondary AS need to be better characterized.

These issues may be addressed with a prospective multi-institutional observational study, through the collection of clinical and pathological data of patients with localized AS.

Involving all reference centres for sarcoma in Italy, the Italian Sarcoma Group (ISG) will be the ideal network for this study, with the collaboration of the Italian Rare Cancer Network (RTR), a 7collaborative network among Italian centres focusing on improving the quality of care of patients with rare tumors.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosis of AS;
* any site of origin;
* any age;
* primary, localized, resectable disease.

Exclusion Criteria: NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * pathological diagnosis of AS;
  * any site of origin;
  * any age;
  * primary, localized, resectable disease.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics | At the time of enrollment
  Demographic data
General characteristics | At the time of enrollment
  Comorbidities
Cancer data | At the time of enrollment
  Previous cancer data
Origin of Tumor | At the time of enrollment
  Site of origin
Tumor characteristics | At the time of enrollment
  Multifocality
Tumor size | At the time of enrollment
  Size
Tumor aspects | 10 years
  Morphological aspects
Pathological characteristics | 10 years
  Proliferative index
Tumor phenotype | 10 years
  Tumor cell phenotype
Molecular characteristics | 10 years
  Molecular aspects

CONTACTS AND LOCATIONS:
Overall Officials: Elena Palassini, Principal Investigator — IRCCS Istituto nazionale Tumori - Milano
Locations (19):
- Italy (19):
  - Istituto Clinico Humanitas Research Hospital IRCCS, Rozzano, Milano
  - Centro Riferimento Oncologico CRO, Aviano, Pordenone
  - AOU San Luigi Gonzaga, Orbassano, Torino
  - Istituto Tumori "Giovanni Paolo II" I.R.C.C.S., Bari
  - Istituto Ortopedico Rizzoli IOR, Bologna
  - Policlinico "Sant'Orsola-Malpighi", Bologna
  - A.O.U. Careggi, Florence
  - Ospedale Policlinico san Martino IRCCS, Genova
  - IRCCS Istituto Nazionale Tumori - Milano, Milan
  - IRCCS Istituto Europeo di Oncologia, Milan
  - Fondazione Irccs San Gerardo Dei Tintori, Monza
  - Istituto Nazionale Tumori_Fondazione "G.Pascale", Napoli
  - IOV Istituto Oncologico Veneto IRCCS, Padua
  - Policlinico "Paolo Giaccone", Palermo
  - Nuovo Ospedale di Prato - S. Stefano, Prato
  - Fondazione Policlinico Campus Biomedico, Roma
  - IRCCS Istituti Fisioterapici Ospitalieri, Roma
  - ASL Ospedale San Giovanni Bosco, Torino
  - Ospedale di Trento, Trento

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Italian Sarcoma Group website — https://www.italiansarcomagroup.org/